CLINICAL TRIAL: NCT00256009
Title: Evacuatio Uteri or Conservtive Treatment After Late Abortion. A Randomize Trial.
Brief Title: Treatment of Late Abortion: Evacuatio Uteri or Conservative Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF 01 279545
Record Dates: First submitted 2005-11-18; First posted 2005-11-21 (Estimated); Last update posted 2006-06-01 (Estimated); Status verified 2005-11

CONDITIONS: Abortion, Spontaneous; Abortion, Induced
Keywords: Late abortion
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Misoprostol

INTERVENTIONS:
Drug: Cytotec

SUMMARY:
A randomize trial: expectation or evacuatio uteri for the treatment after late abortion

DETAILED DESCRIPTION:
A randomize trial adressing 200 women consecutively recruited from clinical practice at Rigshospitalet.Expectation: administration of 800 microgram Cytotec half an hour after delivery. Surgery: Evacuation of the uterus

ELIGIBILITY:
Inclusion Criteria:

abortion at gestational age (ultrasound) 14+0 - 20+0

Exclusion Criteria:

Allergy to cytotec

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200
Dates: Study Completion 2009-01

PRIMARY OUTCOMES:
Side-effect
Complication

SECONDARY OUTCOMES:
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Lars Alling Møller, MD phd, Principal Investigator — Rigshospitalet, Denmark